CLINICAL TRIAL: NCT04521686
Title: A Phase 1 Study of LY3410738 Administered to Patients With Advanced Solid Tumors With IDH1 or IDH2 Mutations
Brief Title: Study of LY3410738 Administered to Patients With Advanced Solid Tumors With IDH1 or IDH2 Mutations
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18077; 2020-002863-77 (EudraCT Number); I9Y-OX-JDHC (Other: Eli Lilly and Company); LOXO-IDH-20002 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma; Chondrosarcoma; Glioma; Any Solid Tumor
Keywords: IDH1; CNS tumor; Cholangiocarcinoma; Chondrosarcoma; Glioma; Glioblastoma; Solid tumor; Primary CNS tumor; Colon cancer; Cancer of the Colon; Colon Neoplasms; Colonic Cancer; Neoplasms, Colonic; Malignant tumor of Breast; Mammary Cancer; Mammary Carcinoma, Human; Mammary Neoplasm, Human; Neoplasms, Breast; Tumors, Breast; Human Mammary Carcinoma; Malignant Neoplasm of Breast; Breast Carcinoma; Breast Tumors; Cancer of the Breast; Breast Neoplasms; Breast Cancer; Thyroid cancer; Prostate cancer; Melanoma; IDH1 R132
MeSH Terms: conditions — Cholangiocarcinoma; Chondrosarcoma; Glioma; Central Nervous System Neoplasms; Glioblastoma; Colonic Neoplasms; Breast Neoplasms; Thyroid Neoplasms; Prostatic Neoplasms; Melanoma | interventions — Gemcitabine; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3410738 (Experimental): Phase 1 dose escalation - Multiple doses of LY3410738
  Interventions: Drug: LY3410738
- LY3410738 alone or in combination with gemcitabine and cisplatin or in combination with durvalumab (Experimental): Phase 1 dose expansion - The maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of LY3410738 alone or in combination with gemcitabine plus cisplatin or in combination with durvalumab
  Interventions: Drug: LY3410738; Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab

INTERVENTIONS:
Drug: LY3410738 — Oral LY3410738
Drug: Gemcitabine — Intravenous gemcitabine
  Other Names: LY188011
  Arms: LY3410738 alone or in combination with gemcitabine and cisplatin or in combination with durvalumab
Drug: Cisplatin — Intravenous cisplatin
  Arms: LY3410738 alone or in combination with gemcitabine and cisplatin or in combination with durvalumab
Drug: Durvalumab — Intravenous durvalumab
  Arms: LY3410738 alone or in combination with gemcitabine and cisplatin or in combination with durvalumab

SUMMARY:
This is an open-label, multicenter Phase 1 study to evaluate safety, tolerability and preliminary efficacy of oral LY3410738 in patients with isocitrate dehydrogenase 1 (IDH1) arginine 132 (R132)-mutant advanced solid tumors, including but not limited to cholangiocarcinoma, chondrosarcoma, and glioma or isocitrate dehydrogenase 2 (IDH2) arginine 140 (R140) or arginine 172 (R172) mutant cholangiocarcinoma.

DETAILED DESCRIPTION:
This is an open-label, multicenter Phase 1 study to evaluate safety, tolerability and preliminary efficacy of oral LY3410738 in patients with IDH1 R132-mutant advanced solid tumors, including but not limited to cholangiocarcinoma, chondrosarcoma, and glioma or IDH2 R140 or R172 mutant cholangiocarcinoma.

This study includes 2 parts: Phase 1 dose escalation and Phase 1 dose expansion. The Phase 1 dose escalation monotherapy cohort will enroll any eligible patient with IDH1 R132-mutant advanced solid tumor or IDH1 or IDH2 mutant cholangiocarcinoma. The Phase 1 dose expansion will include 5 cohorts to further evaluate safety and clinical activity. Three cohorts will be administered LY3410738 monotherapy. The fourth cohort will administer LY3410738 at or below the monotherapy RP2D in combination with gemcitabine and cisplatin. The fifth cohort (US only) will administer LY3410738 at or below the monotherapy RP2D in combination with durvalumab.

IDH1 R132, IDH2 R140, or IDH2 R172 mutations will be identified through genomic testing utilizing material collected prior to patient consent. Molecular assays utilized for enrollment are required to be performed in CLIA, ISO/IEC, CAP, or other similarly certified laboratory. Enrollment of patients with cholangiocarcinoma, chondrosarcoma or glioma may be made based on molecular tests performed in either tumor or blood. Enrollment of patients with other tumor types is limited to testing performed in tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of IDH1 R132 mutation (any solid tumor) or circulating tumor DNA IDH2 R140 or IDH2 R172 mutation (cholangiocarcinoma only) as determined by molecular testing performed at a CLIA, ISO/IEC, CAP, or other similarly certified laboratory. For cholangiocarcinoma, chondrosarcoma, and glioma, molecular testing can be performed on tumor tissue or circulating tumor DNA. For all other solid tumor types, molecular testing must be performed on tumor tissue.
2. Availability of an archived tumor tissue sample. Patients without an available archival tumor tissue sample must be discussed with the sponsor's Medical Monitor prior to enrollment.
3. Eastern Cooperative Oncology Group (ECOG) 0-1.
4. At least 18 years of age.
5. Adequate organ function.
6. Ability to swallow capsules or tablets.
7. Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation.
8. For cholangiocarcinoma patients, must have adequate biliary drainage (per investigator's discretion), with no evidence of ongoing infection.
9. Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and for 3 months following the last dose of study treatment. Patients enrolled to Dose Expansion Cohort 4 shall also follow cisplatin/gemcitabine contraception duration requirements as determined by labels and/or local guidelines. Patients enrolled in dose expansion Cohort 5 should follow durvalumab contraception duration requirements as determined by the durvalumab label and/or local guidelines.

   Monotherapy Dose Escalation:
10. A locally advanced or metastatic solid tumor, where standard curative or palliative measures are no longer effective or are not considered appropriate or safe in the opinion of the investigator.
11. Measurable or non-measurable disease as determined by RECIST 1.1 or RANO as appropriate by tumor type.
12. Prior IDH1 inhibitor treatment is permitted.

    Monotherapy Dose Expansion Cohort 1:
13. Histologically or cytologically confirmed diagnosis of advanced or metastatic cholangiocarcinoma, following 1 to 2 lines of prior systemic treatment for advanced disease. Prior IDH1 inhibitor treatment is not permitted.
14. Measurable disease as determined by RECIST 1.1.

    Monotherapy Dose Expansion Cohort 2:
15. A locally advanced or metastatic solid tumor (except for cholangiocarcinoma), where standard curative or palliative measures are no longer effective or are not considered appropriate or safe in the opinion of the investigator.
16. Measurable disease as determined by RECIST 1.1 or RANO as appropriate by tumor types.

    Monotherapy Dose Expansion Cohort 3:
17. A locally advanced or metastatic solid tumor, where standard curative or palliative measures are no longer effective or are not considered appropriate or safe in the opinion of the investigator.
18. Non-measurable disease only as determined by RECIST 1.1 or RANO as appropriate by tumor type.

    Combination Dose Expansion Cohort 4:
19. Histologically or cytologically confirmed diagnosis of advanced or metastatic cholangiocarcinoma, not eligible for curative resection.
20. No prior systemic therapy for advanced or metastatic disease with the following exceptions:

    * Patients who received adjuvant chemotherapy are eligible, if the adjuvant therapy was completed at least 6 months prior to the development of advanced or metastatic disease.
    * Patients who are receiving up to two cycles of cisplatin plus gemcitabine as the first line systemic therapy while waiting for results of molecule profiling including IDH1/IDH2 mutational status, are eligible, provided that a radiographic assessment during screening demonstrates the absence of interval disease progression since initiation of chemotherapy treatment, and all other eligibility criteria are met.
21. Measurable disease as determined by RECIST 1.1.

    Combination Dose Expansion Cohort 5:
22. Cholangiocarcinoma patients with IDH1 R132, IDH2 R140, or IDH2 R172 mutations
23. Histologically or cytologically confirmed diagnosis of advanced or metastatic cholangiocarcinoma, following 1 or more lines of prior systemic treatment for advanced disease.
24. Measurable disease as determined by RECIST 1.1

Exclusion Criteria:

1. Had an investigational agent or anticancer therapy within 2 weeks; or investigational monoclonal antibody within 4 weeks prior to planned start of LY3410738.
2. Had major surgery within 4 weeks prior to planned start of LY3410738.
3. Had radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of study treatment, except for patients receiving whole brain radiotherapy, which must be completed at least 4 weeks prior to the first dose of study treatment.
4. Patients with cholangiocarcinoma: underwent hepatic radiation, chemoembolization and radiofrequency ablation, radioembolization or other locoregional therapy <4 weeks, have history of hepatic encephalopathy of any grade, have ascites requiring intervention such as diuretics or paracentesis, have ongoing cholangitis, have mixed hepatocellular biliary tract cancer histology or history of liver transplant.
5. Have active CNS metastases are not eligible. Patients with asymptomatic and treated brain metastases may participate provided that they are stable and are not requiring steroid treatment. Patients with suspected or confirmed leptomeningeal disease are not eligible even if treated.
6. Have primary CNS tumors are eligible provided that they do not have leptomeningeal disease and are on a stable or decreasing steroid dose for 7 days prior to screening. Patients with evidence of intracranial hemorrhage either by MRI or CT are not eligible
7. Any unresolved toxicities from prior therapy greater than CTCAE (version 5.0) Grade 2 at the time of starting study treatment except for alopecia.
8. Have clinically significant, uncontrolled cardiac, cardiovascular disease or history of myocardial infarction within 6 months prior to planned start of study treatment.
9. Have active uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator and the sponsor makes it undesirable for the patient to participate in the trial. Screening for chronic conditions is not required.
10. Known active hepatitis B virus (HBV). Note: Controlled (treated) hepatitis will be allowed if they meet the following criteria, antiviral therapy for HBV must be given for at least 1 month prior to first dose of study drug, and HBV viral load must be less than 2000 IU/ml (104 copies/ml) prior to the first dose of study drug. Those on active HBV therapy with viral loads under 2000 IU/ml (104 copies/ml) should stay on the same therapy throughout the study treatment (Appendix E).
11. Known active hepatitis C virus (HCV). Note: Untreated patients with chronic infection by HCV are allowed on study. In addition, successfully treated patients with chronic infection by HCV (defined as sustained virologic response SVR12 or SVR24) are allowed, as long as a minimum of 4 weeks has elapsed between achieving sustained viral response (SVR12 or SVR24) and starting study drug.
12. Known human immunodeficiency virus (HIV); excluded due to potential drug-drug interactions between anti-retroviral medications and LY3410738.
13. Current treatment with certain strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers (Appendix F) and/or P-gp inhibitors (Appendix G).
14. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug.
15. Active second malignancy unless in remission and with life expectancy > 2 years. Refer to protocol exclusion criteria (Section 4.2) for examples of allowed second malignancies.
16. Pregnancy, lactation or plans to breastfeed during the study or within 3 months of the last dose of study intervention.
17. Patients with known hypersensitivity to any component of LY3410738 or its formulation.

    Combination Dose Expansion Cohort 5:
18. Prior treatment with anti-PD 1 or anti-PD L1 therapies.
19. History of Grade 3 or higher immune-related adverse events (irAEs).
20. Active autoimmune disease that has required systemic anti-autoimmune treatment in the past 2 years.

    Endocrine replacement therapy is not considered a form of systemic therapy and is allowed.
21. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids which should not exceed 10 mg/day of prednisone or equivalent corticosteroid.
22. Active interstitial lung disease or history of noninfectious pneumonitis Grade 2 or higher that required treatment with systemic corticosteroids or immunosuppressive drugs.
23. History of hypersensitivity to durvalumab or any excipient.
24. Has received a live vaccine within 30 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 24 months

SECONDARY OUTCOMES:
Objective Response Rate | Up to 24 months
Assess the safety and tolerability of LY3410738 when administered alone or in combination with cisplatin plus gemcitabine or in combination with durvalumab | Up to 24 months
To assess the preliminary anti-tumor activity of LY3410738 when administered alone or in combination with cisplatin plus gemcitabine or in combination with durvalumab | Up to 24 months
Characterize PK properties of LY3410738 when administered alone or in combination with cisplatin plus gemcitabine or in combination with durvalumab | Up to 24 months
To characterize the pharmacodynamic properties of LY3410738 as expressed by change in 2-HG oncometabolite levels in plasma | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (17):
  - Mayo Clinic of Scottsdale, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - USC Norris Cancer Hospital, Los Angeles, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago Pritzker School of Medicine, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- St Vincent's Hospital Sydney, Darlinghurst, New South Wales, Australia
- France (2):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Gustave Roussy, Villejuif
- Prince of Wales Hospital, Hong Kong, Shatin, New Territories, Hong Kong
- Japan (5):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaka University Hospital, Suita-shi, Osaka
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- National University Hospital, Singapore, Singapore
- South Korea (2):
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Seoul National University Hospital, Seoul
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study of LY3410738 in Patients with Advanced Solid Cancer Tumors with a Change in the IDH1 or IDH2 Gene — https://trials.lillytrialguide.com/en-US/trial/1C6aMS1jvpSzT8htklfhXJ?alias=I9Y-OX-JDHC